CLINICAL TRIAL: NCT01270139
Title: Plasmonic Photothermal Therapy of Flow-Limiting Atherosclerotic Lesions With Silica-Gold Nanoparticles: a First-in-Man Study
Brief Title: Plasmonic Nanophotothermal Therapy of Atherosclerosis
Acronym: NANOM-FIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ural State Medical University (Other)
Collaborators: Ural Institute of Cardiology (Other); De Haar Research Task Force (Industry); Ural Federal University (Other); Transfiguration Clinic (Unknown)
Responsible Party: Principal Investigator, Alexander Kharlamov, MD, FESC, FACC, FEACVI, Research manager, De Haar Research Task Force
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NANOM-FIM
Record Dates: First submitted 2010-12-30; First posted 2011-01-05 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Stable Angina; Heart Failure; Atherosclerosis; Multivessel Coronary Artery Disease
Keywords: nanoparticles; mesenchymal stem cell; plasmonics; atherosclerosis; IVUS; stenting
MeSH Terms: conditions — Angina, Stable; Heart Failure; Atherosclerosis | interventions — Stents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nano group (Experimental): 60 patients in Nano group were treated with transplantation of nanoparticles (NP), particularly with a bioengineered patch that was grown with allogenous stem cells pre-cultivated in the medium with NP. After the admission, patients were examined with QCA, and allocated to the trial. The implantation of the patch onto the artery was undergone by the minimally invasive cardiac surgery (MICS CABG) with fixation of the graft to the epicardial myocardium. MICS CABG implies a beating-heart multi-vessel heart surgery performed through several small incisions under direct vision through an anterolateral mini-thoracotomy in the 4th-6th intercostal spaces. The patients can expect high quality of life resuming all everyday activities within a few weeks of their operation. NP were activated with NIR laser at 7 days after the intervention. Patients were treated with bolus of bivalirudin on the day of NP detonation.
  Interventions: Procedure: Transplantation of nanoparticles
- Ferro group (Active Comparator): 60 patients in Ferro group were managed with transplantation of iron-bearing nanoparticles (NP), particularly with intracoronary infusion of allogenous stem cells or CD68 targeted micro-bubbles pre-cultivated in the medium with iron-bearing NP. Cells and/ or micro-bubbles were infused with QCA- and IVUS-guidance to the target coronary artery via micro-catheter on the day of admission. The destruction of CD68 targeted micro-bubbles was obtained by using a Sonos 5500 machine with an S3 transducer operating in ultraharmonic mode (transmit, 1.3MHz/ receive, 3.6 MHz) with a mechanical index of 1.5 and a depth of 4 cm. The AXIOM Artis dBC (Siemens) magnetic navigation system was used for precise delivery of NP to the atheroma through two permanent computer-controlled external magnets generating a navigational magnetic field of 0.08 Tesla in any direction. NP were detonated with NIR laser under the protection of anti-platelet therapy.
  Interventions: Procedure: Transplantation of iron-bearing nanoparticles
- Stenting control (Other): In case of control group (stenting control), XIENCE V stent was implanted to 60 patients. Patients with a single de novo native coronary stenosis of less than 12 mm lesion length, more than 50% stenosis and reference diameter of 3.0 mm as assessed by online QCA were stented by a single stent of 3.0 x 18 mm. The procedure of implantation had to be performed according to common interventional practices including the administration of intracoronary nitroglycerine 0.2 mg of glycerol trinitrate or isosorbide dinitrate and intra-arterial heparin (50-100 U/kg body weight). Predilation with a conventional balloon catheter was recommended before DES deployment according to the manufacturer's recommendation. The protocol recommended the study stent should cover 2 mm of non-diseased tissue on either side of the target lesion. Postdilatation was allowed with a balloon that was shorter than was the study device.
  Interventions: Device: Stenting

INTERVENTIONS:
Procedure: Transplantation of nanoparticles — 60 patients into nanogroup with the use of 60/15-70/40 nm silica-gold nanoparticles (NPs) transplanted by endoscopic cardiac surgery in the composition of bioengineered on-artery patch grown on the basis of biopolymeric scaffold and host circulating CD45-CD34-CD73+CD105+ progenitor cells
  Arms: Nano group
Procedure: Transplantation of iron-bearing nanoparticles — 60 - into ferro-magnetic group with 60/15-70/40 nm silica-gold iron-bearing NPs with delivery in hand of magnetic navigation system
  Arms: Ferro group
Device: Stenting — 60 - in sirolimus-eluting stenting control
  Other Names: XIENCE V
  Arms: Stenting control

SUMMARY:
The investigators hypothesize that the nanoburning is a very challenging technique to demolish and reverse the plaque especially in combination with stem cell technologies promising the functional restoration of the vessel wall.

The completed (in July 2012) interventional three arms (n=180) first-in-man trial (the NANOM-FIM trial) assessed (NCT01270139) the safety and feasibility of two delivery techniques for nanoparticles (NP), and plasmonic photothermal therapy (PPTT) of atherosclerotic lesions. Patients were assigned in a 1:1:1 ratio to receive either (1) nano-intervention with delivery of silica-gold NP in mini-surgery implanted bioengineered on-artery patch (n=60), or (2) nano-intervention with delivery of silica-gold iron-bearing NP with targeted micro-bubbles or stem cells in hands of magnetic navigation system (n=60) versus (3) stent implantation (n=60). The primary outcome was TAV at 12 months.

The observational prospective cohort analysis (an amendment to the protocol of August 29th 2012 with a decision to extend a 1-year study for another 4 years with the assessment of the 5-year clinical outcomes both retro- and prospectively) of the long-term clinical outcomes at the intention-to-treat population of 180 patients with CAD and angiographic SYNTAX score ≤22 enrolled initially to NANOM-FIM trial will be performed at 5 years after the intervention. The primary outcome will be a MACE-free survival. The secondary outcomes will be MACE, cardiac death, TLR (target lesion revascularization) and TVR (target vessel revascularization). Imaging endpoints will be assessed pre-, post- procedure and at 12-month follow-up. Clinical endpoints will be analyzed at the baseline and at 12 and 60-month follow-up (the release of results is expected after October 2016). Parameters of nanotoxicity will be assessed. The independent adjudication analysis of the clinical outcomes is scheduled in 2017-2019.

The subset post-hoc analysis will be conducted at 1- and 5-year follow-up (by the Amendment of August 29th 2012). At the first subset, patients underwent stenting with XIENCE V stent proximal to the site of nano-intervention (n=13). Subjects in the second subset were undergone drug-coated balloon pre-dilation with further nano-technique (n=20). Lesions in patients of the third subset were not prepared for the nano-approach (n=147) (neither stenting nor balloon angioplasty). The analysis will be performed and results will be released after 2018 with the same clinical outcomes.

This project and related manuscripts were not prepared or funded in any part by a commercial organization. Nanoparticles and biomedical equipment were supplied free for the study by the non-profit Agiko and De Haar Research Task Force (Rotterdam-Amsterdam, the Netherlands). All rights of the authors are reserved. The access of the international academic or governmental organizations to the essential and primary data of the trial is restricted by the Russian governmental authorities due to the interest of the Russian Federal Security Service (FSB).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is one of the main cause of disability and death worldwide. The underlying cause generally is atherosclerosis and more in particular thrombotic rupture of an atherosclerotic plaque in a vital artery. The restoration of blood flow to ischemic myocardium is established as the preeminent objective for the treatment of patients with CVD. Some modern angioplasty techniques generally just manipulate the form of the plaque and have some clinical and technical restrictions, relatively high complication rate and restenosis risk.

The most common techniques in current practice are angioplasty with stenting, and CABG surgery (for patients with multivessel disease). Balloon angioplasty and stenting, in fact, manage the form of the plaque and does not create a significant problem of plaque residue flowing from the site. Once a role for elective stent implantation was established, the next goal was to overcome the complications of subacute stent thrombosis (first of all, with the use of drug-eluting stents) and neointimal hyperplasia (bare-metal stents) through pharmacologic and physical means. Among unresolved issues, the investigators can describe restrictions in patients with stenosis of an unprotected left main coronary artery, multivessel disease, diabetes mellitus, still rather high rate of in-stent restenosis, and as a solution of the problem with a foreign body in a vessel, the development of biodegradable stents. Among physical obstacles for stenting, the investigators may note that atherosclerotic plaque build-up can exist in a number of different forms. The plaque can be quite hard and scaly, or more fatty and pliable. Moreover, Dr Peters D. with colleagues from Santa-Barbara (2009) published own data about new modular, multifunctional micelles that contain a targeting element, a fluorophore, and, when desired, a drug component in the same particle. Targeting atherosclerotic plaques in ApoE-KO mice fed a high-fat diet was accomplished with the pentapeptide cysteine-arginine-glutamic acid-lysine-alanine, which binds to clotted plasma proteins. The fluorescent micelles bind to the entire surface of the plaque, and notably, concentrate at the shoulders of the plaque, a location that is prone to rupture. They also show that the targeted micelles deliver an increased concentration of the anticoagulant drug hirulog to the plaque compared with untargeted micelles that may reduce bleeding complications and atherogenesis.

Moreover, the ability of statin drugs to reduce the volume of atherosclerotic plaque in the coronary artery wall, termed plaque regression, has received much attention. The statins have a remarkable track record of lowering cholesterol and improving survival. Apart from lowering low-density lipoprotein cholesterol (LDL-C) levels, they also have a multitude of other actions, often collectively described as pleiotropic effects. JUPITER (2003), REVERSAL (2004), PROVE IT (2004), ESTABLISH (2004), and ASTEROID (2006) trials have shown that low LDL levels after intensive statin therapy when accompanied by raised HDL, can regress, or partially reverse, the plaque buildup in the coronary arteries. The findings suggest that the various components of atheroma respond differently to treatment with medical therapies, and can be used to target plaques that are likely to respond. Thus, lipid pool, inflammatory reaction in the forms of cellular migration, humoral substance release, and oedema are still the most likely to be targets of pharmacotherapy. But, for instance, fibrous tissue, mineral deposits, and ground substance would seem to be irreversible despite metabolic manipulation.

Numerous devices recently have been described that utilize the application of heat to resolve atherosclerotic plaque (laser technique, electrosurgical removing of plaque, or with the use of radio frequency sparking, and others). Plasmonics is a novel invasive approach in medicine, and metal nanoparticles are a new type of optically active composite spherical one consisting of a dielectric core covered by a thin metallic shell which is typically gold. When nanoparticles are irradiated with a near-infrared laser, they absorb energy, which is quickly transferred through nonradiative relaxation into heat and accompanying effects, and eventually leads to irreparable damage of tissue. In oncology, metal nanoparticles may provide a novel means of targeted plasmonic photothermal therapy (PPTT) in tumour tissue, minimizing damage to surrounding healthy tissue. However, this approach does not use in cardiology today possessing the great potential for angioplasty. The efficiency of nanotechnologies, however, is limited by gaps in the current understanding of the thermal interactions between nanoparticles and laser light pulses or continuous waves in the context of complex biological environments. Irradiation, even with moderate pulses of energy, can induce melting, evaporation, and fragmentation of nanoparticles. These events can drastically alter the intended therapeutic effects and lead to the formation of vapour bubbles as well as acoustic waves and shock waves. But the last disadvantages can become advantages depending on the purposes of the treatment. Thus the study opens a new chapter in the history of plasmonics.

The investigators designed this study to check potent clinical opportunities, efficacy and safety of such a novel technique for angioplasty as plasmonic atherodestruction. The investigators have drawn the following research questions: 1) Is it possible to plasmonically entirely destruct a plaque with minimal complications? 2) What level of safety is typical for the different approaches if compare with stenting? 3) What are the advantages and disadvantages of the different delivery techniques - stem cells or magnetic field? 4) What is the meaning of the transplanted mesenchymal CD73+CD105+ stem-progenitor cells for atherosclerosis management? 5) Can plasmonic nanophotothermal therapy (PPTT) get an alternative to stenting?

Plasmonic photothermal therapy (PPTT) can potentially reduce the volume of plaque. PPTT melts an atherosclerotic plaque tissue with irreparable burning of targeted tissues, vapour bubbling of cellular cytoplasm and extracellular matrix with subsequent degradation of tissues, and destructive effects of acoustic and shock waves as the possible plaque-killing mechanisms. NPs are absolutely safe for an organism but entire kinetics is mostly unknown. The most dangerous approach with the lowest level of efficacy and safety is delivery of NPs with microbubbles if compare with stem cell-based one. Mesenchymal stem cells have appropriate effectiveness as a local delivery system with a lot of beneficial properties such as anti-inflammatory, anti-apoptotic, and multi-metabolic effects leading to plaque degradation. Thus, PPTT can become an alternative to stenting.

Among potential problems the investigators may name 1) technique of the delivery of these nanoparticles directly into the plaque (stem cells, aleuronic microbubbles with surfaced antibodies (as a local delivery system), direct injection or infusion into the coronary arteries and plaques during CABG or PCI); 2) high risk of acute fatal atherothrombosis at the heat site due to destruction of the fibrous cap of plaque (role of nanoparticles adhesion on the surface of endothelium); 3) long-term effects of the nanodestruction locally and in entire organism (distribution and effects of accumulation in different organs); 4) mechanism of this effect (plasmonic microexplosion and burning of tissue, lysis of cells due to vapor bubbling of cellular cytoplasm and extracellular tissues, destructive acoustic and shock waves); 5) optimal biophysical parameters and necessary energy levels of nanodetonation to prevent burning of surrounding tissues and perforation of the vessel; 6) plasmonic damage is irreparable, and it means the investigators have to combine it with another biotechnology for the restoration of vessel such as the use of stem cells; 7) optimal type of stem cells (source, origin, level of differentiation, potential, properties).

So, disadvantages of current low-invasive approaches (stenting, statin drugs, and others, laser, electrosurgery devices):

* Foreign body in the heart
* Restenosis, including neointimal hyperplasia (adventitial and circulating stem-progenitor cells of different origin are involved)
* Risk of fatal acute or sub-acute atherothrombosis (including 'in-stent' sub-acute atherothrombosis)
* Non-pathogenetic - cannot reverse or significantly regress the plaque
* No effect for remodeling and calcification (restriction for necessary remodeling)
* Clinical restrictions for some group (multivessel disease, left main CAD, diabetes mellitus, severe CAD and etc), on another hand, CABG is a very traumatic procedure (solution - MICS, including achievements in endoscopic stereotaxic surgery), but CABG is still an approach in charge in severe or high-risk patients

Disadvantages of the studied approach:

* The necessity of the special delivery technique
* The lost function of the artery - irreparable pro-fibrotic damage - the necessity of another clinical management for restoration of tissue - the necessity of the restoration therapy with stem cells
* The threat of acute fatal atherothrombosis due to rupture of (vulnerable) plaque
* Cannot treat non-organic part of plaque - the necessity of the special therapy - stem cells
* The harm of potent detrimental side-effects - vapour bubbling (boiling of cytoplasm and ECM with subsequent lysis of cells, and provocation of pro-apoptotic cascades), acoustic and shock waves due to the plasma-generated laser-related detonation of nanoshells in tissue
* Erratic (uncontrollable) heating - surrounding tissue of the site of interest can achieve a temperature until 38-39°. But at the site of burning final temperature can be at about 50-180 C (cauterization/ searing/ melting effect) with following the pro-fibrous effect of tissue.

ELIGIBILITY:
Inclusion Criteria:

* age 45-65 years old
* male and female
* single- or multi-vessel CAD with flow-limiting lesions
* no indications for coronary artery bypass surgery (CABG)
* stable angina with indications for percutaneous coronary interventions (PCI)
* NYHA (New York Heart Association) I-III functional class of heart failure (HF)
* treated hypertension (in supine position: systole >140 mm Hg, diastole >90 mm Hg)
* de novo treated.

Exclusion Criteria:

* non-compliance,
* angiographic SYNTAX score ≥23
* history of myocardial infarction (MI), unstable angina, PCI or CABG, atrial fibrillation or other dysrhythmias, stroke
* presence of indications for CABG
* presence of contraindications for PCI or CABG
* NYHA IV functional class of HF
* diabetes mellitus (in case of fasting glucose >7.0 mM/L or random glucose >11.0 mM/L)
* untreated hypertension
* asthma
* known hypersensitivity or contraindications to anti-platelet drugs
* contrast sensitivity
* participation to any drug- or intervention-investigation during the previous 60 days

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gabinsky, MD, PhD, DSc, Study Director — Ural Institute of Cardiology; Olga Kovtun, MD, PhD, Study Chair — Ural State Medical University; Alexander Kharlamov, M.D., FESC, FACC, FEACVI, Principal Investigator — De Haar Research Task Force
Locations (4):
- De Haar Research Task Force, Amsterdam, North Holland, Netherlands
- Russia (3):
  - Ural Center of Modern Nanotechnologies, Institute of Natural Sciences, Ural Federal University, Yekaterinburg, Sverdlovsk Oblast
  - Transfiguration Clinic, Yekaterinburg, Sverdlovsk Oblast
  - Ural Institute of Cardiology, Yekaterinburg, Sverdlovsk Oblast

IPD SHARING:
Plan to Share IPD: Yes
The raw data will be partially shared (a Protocol for NANOM-FIM trial and related DREAM project; raw data with atomic force microscopy and scanning electron microscopy) in Mendeley Datasets and ResearchGate without any additional dissemination.
Supporting Information: Study Protocol
Time Frame: The data-sets will be provided in Mendeley and ResearchGate being accompanied to the published articles in 2013-2020.
Access Criteria: There are no specific criteria, but the access to the raw data is partly restricted by the Russian Federal Security Service for indefinite time.
URL: https://doi.org/10.13140/2.1.3109.5847

REFERENCES:
- [Background] Kharlamov AN, Gabinsky JL. Plasmonic photothermic and stem cell therapy of atherosclerotic plaque as a novel nanotool for angioplasty and artery remodeling. Rejuvenation Res. 2012 Apr;15(2):222-30. doi: 10.1089/rej.2011.1305. PMID 22533437
- [Background] Kharlamov AN. Plasmonic photothermal therapy for atheroregression below Glagov threshold. Future Cardiol. 2013 May;9(3):405-25. doi: 10.2217/fca.13.16. PMID 23668744
- [Background] Kharlamov AN. Cardiovascular burden and percutaneous interventions in Russian Federation: systematic epidemiological update. Cardiovasc Diagn Ther. 2017 Feb;7(1):60-84. doi: 10.21037/cdt.2016.08.10. PMID 28164014
- [Background] Kharlamov AN. Glimpse into the Future of Nanotheranostic Strategies for Regression of Atherosclerosis through the Prism of Systems Biomedicine: Systematic Review of Innovations from Multifunctional Nanoformulations to Devices on Chip. Current Nanomedicine 6(3): 186-218, 2016. doi: 10.2174/2468187306666161121142756.
- [Background] Kharlamov AN, Zubarev IV, Shishkina EV, Shur VY. Nanoparticles for treatment of atherosclerosis: challenges of plasmonic photothermal therapy in translational studies. Future Cardiol. 2018 Mar;14(2):109-114. doi: 10.2217/fca-2017-0051. Epub 2018 Jan 16. No abstract available. PMID 29336170
- [Result] Kharlamov AN, Tyurnina AE, Veselova VS, Kovtun OP, Shur VY, Gabinsky JL. Silica-gold nanoparticles for atheroprotective management of plaques: results of the NANOM-FIM trial. Nanoscale. 2015 May 7;7(17):8003-15. doi: 10.1039/c5nr01050k. PMID 25864858
- [Result] Kharlamov AN, Feinstein JA, Cramer JA, Boothroyd JA, Shishkina EV, Shur V. Plasmonic photothermal therapy of atherosclerosis with nanoparticles: long-term outcomes and safety in NANOM-FIM trial. Future Cardiol. 2017 Jul;13(4):345-363. doi: 10.2217/fca-2017-0009. Epub 2017 Jun 23. PMID 28644056
- See also: Ural Institute of Cardiology — http://www.cardio-burg.ru
- See also: Ural Center of Modern Nanotechnologies, Institute of Natural Sciences, Ural Federal University — http://nanocenter.urfu.ru/en
- See also: Transfiguration Clinic — http://www.pr-clinica.ru
- See also: De Haar Research Task Force — https://www.dhrfpro.com/
- Available data/document: Study Protocol: doi: 10.13140/2.1.3109.5847 — https://www.researchgate.net/publication/273623828_Protocol_v31_of_NANOM-FIM_trial — The protocol of the trial (v. 3.1.) was released in ResearchGate in March 2015.
- Available data/document: Study Protocol: doi: 10.17632/rkz98ttjrd.1 — https://data.mendeley.com/datasets/rkz98ttjrd/1 — This is a protocol of NANOM-FIM trial released in Mendeley Datasets.
- Available data/document: Individual Participant Data Set: doi: 10.17632/5hzb3249hn.1 — https://data.mendeley.com/datasets/5hzb3249hn/1 — There is Atomic Force Microscopy data from random patients.
- Available data/document: Protocol and Proposal of the Research Project: doi: 10.13140/RG.2.1.4913 — https://www.researchgate.net/publication/286927115_Development_of_bioresorbable_scaffolds_and_nanotechnologies_for_reversal_of_atherosclerosis_DREAM — This is a set of documents of the related DREAM project funded by the FP7/ European Commission. The DREAM study was a collaborative project at the loop between Erasmus MC (Rotterdam, The Netherlands) and Ural Institute of Cardiology (Yekaterinburg, Russia) including NANOM-FIM trial.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was a multi-centre (two sites), observational, open-label, three arms study in 180 patients with CAD and angiographic SYNTAX score ≤22. The project started in April, 2007 and completed in June, 2012.
Pre-assignment Details: Some patients were excluded from the per-treatment-evaluable population since they received a stent or were treated with CABG as an event of target lesion revascularization (TLR). Patients were also excluded in case of non-compliance or documented while the ongoing trial the first arose diabetes, NYHA IV functional class of HF, or SYNTAX score ≥23.
Groups:
- Nano Group: 60 patients in Nano group were treated with bioengineered patch that was grown with allogeneic stem cells pre-cultivated in the medium with NP. After the admission, patients were examined with QCA, and allocated to the trial. The implantation of the patch onto the artery was undergone by the minimally invasive cardiac surgery (MICS CABG) with fixation of the graft to the epicardial myocardium. MICS CABG implies a beating-heart multi-vessel heart surgery performed through several small incisions under direct vision through an anterolateral mini-thoracotomy in the 4th-6th intercostal spaces. The approach considered as an alternative to PCI allowing quick recover without major complications. The patients can expect high quality of life resuming all everyday activities within a few weeks of their operation. NP were activated with NIR laser at 7 days after the intervention. Patients were treated with bolus of bivalirudin on the day of NP detonation.
- Ferro Group: 60 patients in Ferro group were managed with intracoronary infusion of allogeneic stem cells or CD68 targeted micro-bubbles pre-cultivated in the medium with iron-bearing NP. Cells and/ or micro-bubbles were infused with QCA- and IVUS-guidance to the target coronary artery via micro-catheter on the day of admission at the Acute Care Unit. The destruction of CD68 targeted micro-bubbles was obtained by using a Sonos 5500 machine with an S3 transducer operating in ultraharmonic mode (transmit, 1.3MHz/ receive, 3.6 MHz) with a mechanical index of 1.5 and a depth of 4 cm. The AXIOM Artis dBC (Siemens) magnetic navigation system was used for precise delivery of NP to the atheroma through two permanent computer-controlled external magnets generating a navigational magnetic field of 0.08 Tesla in any direction with opportunity to produce a spot at the area of target artery and lesion. NP were detonated with NIR laser at the end of the procedure under the protection of anti-platelet therapy.
- Stenting Control: In case of control group, XIENCE V stent was implanted to 60 patients. Patients with a single de novo native coronary stenosis of less than 12 mm lesion length, more than 50% stenosis and reference diameter of 3.0 mm as assessed by online QCA were stented by a single stent of 3.0 x 18 mm. The procedure of implantation had to be performed according to common interventional practices including the administration of intracoronary nitroglycerine 0.2 mg of glycerol trinitrate or isosorbide dinitrate and intra-arterial heparin (50-100 U/kg body weight). Predilation with a conventional balloon catheter was recommended before DES deployment according to the manufacturer's recommendation. The protocol recommended the study stent should cover 2 mm of non-diseased tissue on either side of the target lesion. Postdilatation was allowed with a balloon that was shorter than was the study device.
Period: Overall Study
Arm/Group | Nano Group | Ferro Group | Stenting Control
Started | 60 (Intention-to-treat population) | 60 (Intention-to-treat population) | 60 (Intention-to-treat population)
Completed | 42 (Pre-treatment evaluable population) | 34 (Pre-treatment evaluable population) | 40 (Pre-treatment evaluable population)
Not Completed | 18 | 26 | 20
Not completed — Adverse Event | 8 | 17 | 18
Not completed — Lost to Follow-up | 10 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nano Group | Ferro Group | Stenting Control | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 60 | 180
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (10.3) | 50.9 (8.8) | 52.6 (6.8) | 51.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 14 | 41
  Male | 49 | 44 | 46 | 139
Region of Enrollment [Number; unit: participants]
  Russian Federation | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Total Atheroma Volume
Description: Total atheroma volume (TAV, plaque-media volume, mm3) at 12 months. Quantitative coronary angiography (QCA) and Intravascular Ultrasound (IVUS) were performed pre-, post-procedure and at 12-month follow-up after a bolus infusion of i.c. nitrate. QCA was undergone with the CAAS II analysis system (Pie Medical B.V., Maastricht, The Netherlands) with analysis of different QCA parameters such as minimal lumen diameter, maximum lumen diameter, reference diameter, diameter stenosis, lesion length, percent atheroma volume (PAV), total atheroma volume (TAV), and lumen volume.
Time Frame: at 12-month follow-up
Population: The intention-to-treat-population analysis
Measure: Mean (Standard Deviation); unit: mm3
Groups:
- Nano Group: 60 patients in Nano group were treated with bioengineered patch that was grown with allogenous stem cells pre-cultivated in the medium with NP. After the admission, patients were examined with QCA, and allocated to the trial. The implantation of the patch onto the artery was undergone by the minimally invasive cardiac surgery (MICS CABG) with fixation of the graft to the epicardial myocardium. MICS CABG implies a beating-heart multi-vessel heart surgery performed through several small incisions under direct vision through an anterolateral mini-thoracotomy in the 4th-6th intercostal spaces. The approach considered as an alternative to PCI allowing quick recover without major complications. The patients can expect high quality of life resuming all everyday activities within a few weeks of their operation. NP were activated with NIR laser at 7 days after the intervention. Patients were treated with bolus of bivalirudin on the day of NP detonation.
- Ferro Group: 60 patients in Ferro group were managed with intracoronary infusion of allogenous stem cells or CD68 targeted micro-bubbles pre-cultivated in the medium with iron-bearing NP. Cells and/ or micro-bubbles were infused with QCA- and IVUS-guidance to the target coronary artery via micro-catheter on the day of admission at the Acute Care Unit. The destruction of CD68 targeted micro-bubbles was obtained by using a Sonos 5500 machine with an S3 transducer operating in ultraharmonic mode (transmit, 1.3MHz/ receive, 3.6 MHz) with a mechanical index of 1.5 and a depth of 4 cm. The AXIOM Artis dBC (Siemens) magnetic navigation system was used for precise delivery of NP to the atheroma through two permanent computer-controlled external magnets generating a navigational magnetic field of 0.08 Tesla in any direction with opportunity to produce a spot at the area of target artery and lesion. NP were detonated with NIR laser at the end of the procedure under the protection of anti-platelet therapy.
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
mm3 | 108.2 (42.2) | 115.6 (64) | 178 (52.6)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis - Nano group is superior to Ferro group and stenting control; Test type: Non-Inferiority or Equivalence — The sample size was not defined on the basis of an end-point hypothesis, therefore the present FIM study should be considered as hypothesis-generating; p < 0.05, ANOVA — Overall comparison was assessed by applying the Friedman test, and pairwise comparisons between post-procedure and follow-up (nano vs ferro, nano vs stenting, and ferro vs stenting) were performed by ANOVA

2. Primary Outcome: MACE (Major Adverse Cardiovascular Events)-Free Survival
Description: MACE (major adverse cardiovascular events)-free survival reflects per cent of survived patients without MACE. An amendment to the protocol was approved on August 29th 2012 with a decision to extend a 1-year study for another 4 years with the assessment of the 5-year clinical outcomes both retro- and prospectively.
Time Frame: at 60 months follow-up
Population: Some patients were lost to follow-up at 5 years and were not included to the final analysis. The intention-to-treat analysis was performed at 60 months.
Measure: Number; unit: Percentage of survivors without MACE
Groups:
- Nano Group: 60 patients in Nano group were treated with transplantation of nanoparticles (NP), particularly with a bioengineered patch that was grown with allogenous stem cells pre-cultivated in the medium with NP. After the admission, patients were examined with QCA, and allocated to the trial. The implantation of the patch onto the artery was undergone by the minimally invasive cardiac surgery (MICS CABG) with fixation of the graft to the epicardial myocardium. MICS CABG implies a beating-heart multi-vessel heart surgery performed through several small incisions under direct vision through an anterolateral mini-thoracotomy in the 4th-6th intercostal spaces. The patients can expect high quality of life resuming all everyday activities within a few weeks of their operation. NP were activated with NIR laser at 7 days after the intervention. Patients were treated with bolus of bivalirudin on the day of NP detonation. Transplantation of nanoparticles: 60 patients into nanogroup with the use of 60/
- Ferro Group: 60 patients in Ferro group were managed with transplantation of iron-bearing nanoparticles (NP), particularly with intracoronary infusion of allogenous stem cells or CD68 targeted micro-bubbles pre-cultivated in the medium with iron-bearing NP. The destruction of CD68 targeted micro-bubbles was obtained by using a Sonos 5500 machine with an S3 transducer operating in ultraharmonic mode (transmit, 1.3MHz/ receive, 3.6 MHz) with a mechanical index of 1.5 and a depth of 4 cm. The AXIOM Artis dBC (Siemens) magnetic navigation system was used for precise delivery of NP. NP were detonated with NIR laser under the protection of anti-platelet therapy. Transplantation of iron-bearing nanoparticles: 60 - int
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of survivors without MACE | 94.3 | 91.4 | 90.5
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Other — The Kolmogorov-Smirnov test was used to prove Gaussian distribution allowing for calculation of the mean and standard deviation. Non-Gaussian samples are described by median and range. Discriminant variables are evaluated with the two-sided Fisher's exact test. Differences between three groups were analyzed by means of a repeated-measures oneway ANOVA followed by a Fisher's post hoc test. We used the Cox proportional hazards ratios (HR) and 95% CI for the end points; p < 0.05, Kaplan-Meier — A p value was calculated for each comparison separately, and indicated as "for all comparisons". In case if p value was >0.05, it was mentioned with a separated info. The threshold for statistical significance was a p value below 0.05

3. Secondary Outcome: Per Cent of Fibro-fatty Component
Description: IVUS (intravascular ultrasound) and IVUS-VH (virtual histology) images were acquired simultaneously with a phased array 20 MHz intravascular ultrasound catheter EagleEye (Volcano Co., Rancho Cordova, CA, USA) with motorized pull-back at a constant speed of 0.5 mm/s. Four tissue components (necrotic core - red; dense calcium - white; fibrous - green; and fibro-fatty - light green or yellow) were identified with autoregressive classification systems. For each cross section stent struts were detected as areas of apparent dense calcium and necrotic core. All IVUS analysis was performed offline by a CoreLab of the Ural Institute of Cardiology.
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: Percentage of tissue
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of tissue | 16.06 (8.53) | 16.46 (8.15) | 11.32 (3.84)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis - Nano group is superior to Ferro group and stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Event Free Survival
Description: The Kaplan-Meier analysis of the cardiac event-free survival (failure-free survival). The end point in this study was cardiac event-free survival during follow-up, starting at randomization. Cardiac events included cardiac death, myocardial infarction and unintended revascularization. Cardiac death was defined as sudden death, death after the onset of symptoms suggestive of cardiac ischemia and death due to heart failure. Noncardiac death was defined as death due to all other causes. Myocardial infarction was defined as an increase in cardiac enzymes or new pathologic Q-waves on the ECG, or both. Unintended revascularization was defined as PTCA or CABG performed due to worsening of the patient's clinical condition, rather than the PTCA or CABG assigned by the revascularization team when patient management was determined.
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Number; unit: Percentage of survived patients
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of survived patients | 91.7 | 81.7 | 80
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, Kaplan-Meier

5. Secondary Outcome: Restenosis Rate
Description: Restenosis (stenosis>50%) rate
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Number; unit: Percentage of patients
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of patients | 3.33 | 3.33 | 10
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nano group is superior to Ferro group and Stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, Chi-squared

6. Secondary Outcome: Late Definite Thrombosis
Description: Late definite thrombosis rate
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of participants | 0 | 1.7 | 6.7
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nano group is superior to Ferro group and Stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, Chi-squared

7. Secondary Outcome: Coronary Vasomotion - Mean Lumen Diameter After Infusion of Acetylcholine 10-6 M
Description: Coronary vasomotion was assessed with QCA. End-diastolic images of coronary arteries were evaluated at baseline, after intravascular infusion of acetylcholine (through a microcatheter at increasing doses up to 10-8, 10-7, 10-6 M with a washout period of at least five minutes between each dose), and after nitroglycerine application following acetylcholine (100 µg orally). In all patients, measurements were performed in two segments on site of intervention while 960 seconds. The artery diameter was calibrated against the contrast-filled tip of the catheter. Vasoconstriction to acetylcholine was defined as a 3% change of the mean lumen diameter after infusion of the maximal dose of acetylcholine. An investigator blinded to treatment group performed all measurements.
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
mm | 4.15 (0.34) | 3.91 (0.55) | 2.88 (0.69)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Per Cent Atheroma Volume
Description: Per cent atheroma volume (PAV, plaque burden, %). Quantitative coronary angiography (QCA) and Intravascular Ultrasound (IVUS) were performed pre-, post-procedure and at 12-month follow-up after a bolus infusion of i.c. nitrate. QCA was undergone with the CAAS II analysis system (Pie Medical B.V., Maastricht, The Netherlands) with analysis of different QCA parameters such as minimal lumen diameter, maximum lumen diameter, reference diameter, diameter stenosis, lesion length, percent atheroma volume (PAV), total atheroma volume (TAV), and lumen volume.
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: Percentage of tissue
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of tissue | 37.8 (13.9) | 39.4 (12.8) | 52.9 (15.8)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nanogroup is superior to Ferro group and stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Target Lesion Revascularization
Description: Target lesion revascularization, per cent
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of participants | 3.3 | 3.3 | 6.7
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nanogroup is superior to Ferro group and stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, Chi-squared

10. Secondary Outcome: Per Cent of Fibrous Component
Description: as for outcome 3
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: Percentage of tissue
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of tissue | 48.81 (12.96) | 50.95 (12.04) | 60.38 (9.92)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Per Cent of Necrotic Core
Description: as for outcome 3
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: Percentage of tissue
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of tissue | 28.47 (9.53) | 26.58 (9.36) | 25.47 (10.05)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nano groups is superior to Ferro group and Stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Per Cent of Calcium
Description: as for outcome 3
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: Percentage of tissue
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of tissue | 6.57 (1.92) | 6.01 (1.85) | 2.83 (1.69)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nano group is superior to Ferro group and Stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Minimal Lumen Diameter
Description: Minimal lumen diameter (MLD, mm)
Time Frame: at 12-month follow-up
Population: The intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
mm | 3.08 (0.52) | 2.98 (0.63) | 2.82 (0.32)
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; The null hypothesis is Nano groups is superior to Ferro group and Stenting control; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]

14. Secondary Outcome: MACE
Description: MACE includes per cent of patients with cardiac death. STEMI (ST-elevation myocardial infarction), non-STEMI, and TLR (target lesion revascularization). An amendment to the protocol was approved on August 29th 2012 with a decision to extend a 1-year study for another 4 years with the assessment of the 5-year clinical outcomes both retro- and prospectively.
Time Frame: at 60 months follow-up
Population: The intention-to-treat analysis was performed at 60 months.
Measure: Number; unit: Percentage of participants with MACE
Groups:
- Nano Group: 60 patients in Nano group were treated with transplantation of nanoparticles (NP), particularly with a bioengineered patch that was grown with allogenous stem cells pre-cultivated in the medium with NP. The implantation of the patch onto the artery was undergone by the minimally invasive cardiac surgery (MICS CABG) with fixation of the graft to the epicardial myocardium. MICS CABG implies a beating-heart multi-vessel heart surgery performed through several small incisions under direct vision through an anterolateral mini-thoracotomy in the 4th-6th intercostal spaces. NP were activated with NIR laser at 7 days after the intervention. Transplantation of nanoparticles: 60 patients into nanogroup with the use of 60/15-70/40 nm silica-gold nanoparticles (NPs) transplanted by endoscopic cardiac surgery in the composition of bioengineered on-artery patch grown on the basis of biopolymeric scaffold and host circulating CD45-CD34-CD73+CD105+ progenitor cells
- Ferro Group: 60 patients in Ferro group were managed with transplantation of iron-bearing nanoparticles (NP), particularly with intracoronary infusion of allogenous stem cells or CD68 targeted micro-bubbles pre-cultivated in the medium with iron-bearing NP. The destruction of CD68 targeted micro-bubbles was obtained by using a Sonos 5500 machine with an S3 transducer operating in ultraharmonic mode (transmit, 1.3MHz/ receive, 3.6 MHz) with a mechanical index of 1.5 and a depth of 4 cm. The AXIOM Artis dBC (Siemens) magnetic navigation system was used for precise delivery of NP to the atheroma through two permanent computer-controlled external magnets generating a navigational magnetic field of 0.08 Tesla in any direction. NP were detonated with NIR laser under the protection of anti-platelet therapy.
  Transplantation of iron-bearing nanoparticles: 60 - into ferro-magnetic group with 60/15-70/40 nm silica-gold iron-bearing NPs with delivery in hand of magnetic navigation system
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 60 | 60 | 60
Percentage of participants with MACE | 14.3 | 20.9 | 22.9
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.05, Kaplan-Meier — [p-value comment as in outcome 2, analysis 1]

15. Secondary Outcome: Cardiac Death
Description: Cardiac death includes per cent of patients passed away due to any cardiac death. An amendment to the protocol was approved on August 29th 2012 with a decision to extend a 1-year study for another 4 years with the assessment of the 5-year clinical outcomes both retro- and prospectively.
Time Frame: at 60 months follow-up
Population: The per-treatment-evaluable analysis was performed at 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 47 | 51 | 51
Participants | 2 | 3 | 3
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.05, Kaplan-Meier — [p-value comment as in outcome 2, analysis 1]

16. Secondary Outcome: TLR (Target Lesion Revascularization)
Description: TLR (target lesion revascularization) reflects per cent of patients with TLR. An amendment to the protocol was approved on August 29th 2012 with a decision to extend a 1-year study for another 4 years with the assessment of the 5-year clinical outcomes both retro- and prospectively.
Time Frame: at 60 months follow-up
Population: The per-treatment-evaluable analysis was performed at 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 47 | 51 | 51
Participants | 4 | 5 | 6
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.05, Kaplan-Meier — [p-value comment as in outcome 2, analysis 1]

17. Secondary Outcome: TVR (Target Vessel Revascularization)
Description: TVR (target vessel revascularization) reflects per cent of patients with TVR. An amendment to the protocol was approved on August 29th 2012 with a decision to extend a 1-year study for another 4 years with the assessment of the 5-year clinical outcomes both retro- and prospectively.
Time Frame: at 60 months follow-up
Population: The per-treatment-evaluable analysis was performed at 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Nano Group | Ferro Group | Stenting Control
Number analyzed (Participants) | 47 | 51 | 51
Participants | 10 | 16 | 14
Statistical Analysis 1: Comparison: Nano Group vs Ferro Group vs Stenting Control; Null hypothesis is Nano group is superior to Ferro group and stenting control; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.05, Kaplan-Meier — [p-value comment as in outcome 2, analysis 1]

18. Secondary Outcome: Mean Number of Membrane Defects on Membrane of Red Blood Cells
Description: Mean number of membrane defects on membrane of red blood cells calculated with atomic force microscopy (AFM) in random patients. An amendment to the protocol was approved on August 29th 2012 with a decision to extend a 1-year study for another 4 years with the assessment of the 5-year clinical outcomes both retro- and prospectively.
Time Frame: at 60 months follow-up
Population: The analysis was undergone in eligible random evaluable patients. Only one random patient with exposure of gold nanoparticles was selected for a trial-balloon analysis of cytotoxicity. The blood was collected and split blindly into two ex-vivo experiments with AFM microscopy (see description).
Measure: Number; unit: Mean number of membrane defects per cell
Units Other Than Participants: Area of blood sample per patient
Groups:
- Exposure of Nanoparticles: Blood for ex-vivo cytotoxic analysis (20.0 ml from a random patient) was collected for analysis at the Center for Modern Nanotechnologies of the Ural Federal University from the random naive patients to the BD Vacutainer (NJ, USA) plastic heparin tubes (spray-coated) with 150 USP units of sodium heparin per 10.0 ml, and then diluted by 0.1 g/l silica-gold NPs.
- Sham: Blood for ex-vivo cytotoxic analysis (20.0 ml from a random patient) was collected for analysis at the Center for Modern Nanotechnologies of the Ural Federal University from the random naive patients to the BD Vacutainer (NJ, USA) plastic heparin tubes (spray-coated) with 150 USP units of sodium heparin per 10.0 ml, and then diluted by saline.
Arm/Group | Exposure of Nanoparticles | Sham
Number analyzed (Participants) | 1 | 1
Number analyzed (Area of blood sample per patient) | 5 | 5
Mean number of membrane defects per cell | 6.12 | 1.12
Statistical Analysis 1: Comparison: Exposure of Nanoparticles vs Sham; Null hypothesis is ex-vivo arm with exposure of nanoparticles is superior to saline control; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Only parameters related to event free survival were assessed in patients who have completed the trial with the final follow-up. Some patients were excluded (64/180, a 35.6% of the intention-to-treat population) during the trial due to non-compliance, broken randomization codes or violations of the protocol.
Arm/Group | Nano Group | Ferro Group | Stenting Control
All-Cause Mortality (participants affected / at risk) | 5/42 | 11/34 | 12/40
Serious Adverse Events (participants affected / at risk) | 8/42 | 17/34 | 18/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/34 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nano Group (N=42) | Ferro Group (N=34) | Stenting Control (N=40)
Target lesion cardiac death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Cardiac death which is related to the intervention at the site of target lesion
Target vessel cardiac death (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) — Cardiac death which is not related to the intervention at the target lesion
Non-cardiac death (Vascular disorders) | 5 (5) | 9 (9) | 10 (10) — Death due to stroke, cancer, trauma and others
Target lesion myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) — Myocardial infarction which is related to the intervention at the target lesion
Target vessel myocardial infarction (Cardiac disorders) | 3 (3) | 6 (6) | 4 (4) — Myocardial infarction which is not related to the intervention at the target lesion

LIMITATIONS AND CAVEATS:
The study was launched as a PROBE trial. But randomization was broken because of the specific study design, where procedures differ significantly, and impossibility to calculate sample size due to absolute novelty of the technology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This project and manuscript were not prepared or funded in any part by a commercial organization. Nanoparticles and biomedical facilities were supplied free for the study by the non-profit Agiko Foundation (Yekaterinburg, Russia). All rights of authors are reserved by the Russian Law. The access of the non-russian international and alien academic and governmental organizations to the essential and primary documents of the trial is restricted by the Russian government.